CLINICAL TRIAL: NCT03913247
Title: Evaluation of Methods for Extrapolating or Estimating the Size of Children in Pediatric Intensive Care Compared With the Reference Method of the World Health Organization (WHO)
Brief Title: Evaluation of Methods for Extrapolating or Estimating the Size of Children in Pediatric Intensive Care
Acronym: EvTaReaP
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0031
Record Dates: First submitted 2019-04-10; First posted 2019-04-12 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group with different size measures: Each patient included in the study will have different measure of size.
  Interventions: Other: Size Measurement using a measuring tape, a caliper and a metric

INTERVENTIONS:
Other: Size Measurement using a measuring tape, a caliper and a metric — Each patient will have the following measure: measure of the span, the tibia, the ulna, the distance between the hill and the knee, the head, the trunk and the leg. The different measures will be done using a measuring tape and with a caliper. Before leaving the intensive care unit, each patients will be measured according to the WHO standard, that is to say strictly lengthened, using a metric for patient younger than 2 and stand up using a stadiometer for patient older than 2.

SUMMARY:
Size is a key data used daily by dietary teams; the paramedical team, nurse and diet are in charge of its measures.

In pediatric intensive care unit, a reliable size of the child must be obtained. It allows to realize:

* a nutritional assessment based on the World Health Organization (WHO) nutritional indices such as the Body Mass Index (BMI), growth chart monitoring and other nutritional indices. Nutritional status should be assessed and followed in pediatric intensive care as it is correlated with the prognosis of children.
* an estimate of the energy needs by calculation of the rest energy expenditure.
* a calculation of the body surface, useful for drug prescription, evaluation of burn scores, calculation of water and energy requirements and indexing of hemodynamic and ventilatory data.

An error in size measurement results in an error in BMI, calculation of energy requirements, and body surface area.

The WHO has defined "gold standard" criteria for measuring height in children, distinguishing the less than two years in whom the size is measured strictly lengthened, using a metric, and the more than two years in which height is measured standing with a stadiometer. In the context of pediatric resuscitation, the criteria for WHO size measurement are difficult to meet (coma, sedation, respiratory assistance, catheter, monitoring, proclive position, etc.) compromising standing or rectitude required for measurements.

The child is a growing organism. Health book sizes and declarative sizes are not always up-to-date.

It is therefore important to overcome these difficulties by using estimating or extrapolation methods that are applicable and safe in pediatric intensive care unit.

Currently, in pediatric intensive care units, the size evaluation, by direct measurement, estimation or extrapolation of segmental measurement, is not systematic because of the complexity of the measurement; To date, no method is used as a reference method in pediatric intensive care.

Among Children in pediatric intensive care unit (which does not usually meet the criteria of the WHO Gold Standard for Measurement of Height), to determine the optimal method for size measurement, by comparing different methods of estimating / extrapolating the size, gold standard WHO (achievable after the stay in intensive care).

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 28 days to 18 years old.
* Admitted in pediatric intensive care unit with a resuscitation situation (at least one system failure including respiratory and/or hemodynamic and/or neurological).
* Children whose size was not measurable, at the time of the admission in pediatric intensive care unit according to WHO standards.
* Patient affiliated to a social security system

Exclusion Criteria:

* No expected evolution to a clinical state allowing the size measure according to the WHO standards according to age.
* Stature growth greater (defined by WHO growth velocity scale according to age and sex) than 5% before the expected delay allowing the size measure using the WHO standards according to age
* Children with skeleton malformation, dwarfism, abnormal limb.
* Expected death before the end of the stay in pediatric intensive care unit
* Parents or patients able to answer, refusing to participate to the study

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients in pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 477 (Actual)
Dates: Start 2019-11-29 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-26 (Actual)

PRIMARY OUTCOMES:
reliability of a series of extrapolation measurement techniques or size estimation in pediatric intensive care units. | 150 days
  The reliability of the estimation / size extrapolation methods will be defined by the average relative error relative to the WHO gold standard. A method will be considered reliable and without clinical impact if the absolute value of the average relative error is less than 3.5%

CONTACTS AND LOCATIONS:
Overall Officials: Carole Ford-Chessel, Principal Investigator — Hospices Civils de Lyon
Locations (10):
- Service de réanimation pédiatrique Hôpital Reine Fabiola Hôpital Publique, Brussels, Belgium
- France (7):
  - Service de réanimation pédiatrique Centre hospitalier universitaire de Bordeaux, Bordeaux
  - Hôpital Femme Mère Enfant, Bron
  - Service de réanimation pédiatrique Hôpital cardiologique Louis Pradel, Bron
  - Service de réanimation et de surveillance continue pédiatrique CHRU de Lille, Lille
  - Service de réanimation pédiatrique CHU La Timone AP-HM, Marseille
  - Service de réanimation pédiatrique Centre hospitalier universitaire de Nantes, Nantes
  - Service de réanimation pédiatrique Rue Du Morvan (CHRU NANCY - HOPITAUX DE BRABOIS), Vandœuvre-lès-Nancy
- Service de réanimation pédiatrique Hôpital de l'hôtel dieu de France, Beirut, Lebanon
- Haute école de santé - HES-SO Genève, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ford Chessel C, Berthiller J, Haran I, Tume LN, Bourgeaud C, Tsapis M, Gaillard-Le Roux B, Gauvard E, Loire C, Guillot C, Mouneydier K, Nolent P, Blache T, Cour Andlauer F, Rooze S, Jotterand Chaparro C, Morice C, Subtil F, Huot M, Valla FV. Accurate height and length estimation in hospitalized children not fulfilling WHO criteria for standard measurement: a multicenter prospective study. Eur J Pediatr. 2024 Oct;183(10):4275-4286. doi: 10.1007/s00431-024-05692-3. Epub 2024 Jul 25. PMID 39052138